CLINICAL TRIAL: NCT01545804
Title: Lenalidomide as Second-line Treatment for Advanced Hepatocellular Carcinoma (HCC): a Phase II Clinical Trial
Brief Title: Lenalidomide as Second-line Treatment for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201105063MB
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Liver Cancer
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — All enrolled patients will receive Lenalidomide, 25 mg orally daily, until objective disease progression, development of unacceptable toxicity, or voluntary discontinuation by the subjects.

SUMMARY:
This is a single-arm, open-label phase II trial. Eligible patients must have histological or clinical diagnosis of Hepatocellular Carcinoma (HCC), advanced tumors that are not amenable to loco-regional therapy, documented progression with or intolerance to sorafenib-based treatment or other anti-angiogenic therapy as first-line therapy for advanced HCC.

DETAILED DESCRIPTION:
This is a single-arm, open-label phase II trial. Eligible patients must have histological or clinical diagnosis of HCC, advanced tumors that are not amenable to loco-regional therapy, documented progression with or intolerance to sorafenib-based treatment or other anti-angiogenic therapy as first-line therapy for advanced HCC, ECOG performance status 0 or 1, Child-Pugh class A liver function, and measurable tumors (by RECIST 1.1). All enrolled patients will receive lenalidomide, starting at 25 mg orally daily on days 1-21, every 4 weeks. Lenalidomide treatment will continue until objective disease progression, development of unacceptable toxicity, or voluntary discontinuation. Dose titration will be done according to the severity of adverse events. Tumor assessment will be done after 4 weeks and 8 weeks of treatment and every 8 weeks thereafter until objective disease progression. All patients will receive DCE-MRI at baseline, on day 3 ± 1 day, and on day 14 ± 2 days. The primary endpoint is the percentage of patients who are tumor progression-free (according to RECIST 1.1) at 6 months after lenalidomide treatment. It is estimated that in the 2nd-line setting, 20% or less patients will remain progression-free at 6 months with current treatment, i.e., no standard treatment. Lenalidomide will be considered effective if the percentage of patients who remain progression-free at 6 months can be increased to 40%. With type I and type II errors of 0.05 and 0.1, respectively, 50 evaluable patients, i.e., patients who receive at least 4 weeks of study medication and receive the first scheduled assessment of tumor response, will be required and the planned sample size will be 55 patients, assuming a 10% dropout rate. The study is expected to complete in 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed HCC, OR clinically diagnosed HCC
* Documented progression with or intolerance to first-line molecular targeted therapy as first-line therapy for advanced HCC.
* Acceptable first-line molecular targeted therapies include (1) sorafenib monotherapy and sorafenib-based combination; (2) anti-angiogenic therapy including brivanib, linifanib, pazopanib, bevacizumab, dovitinib (TKI258), and vargatef (BIBF1120).
* For patients who receive first-line sorafenib monotherapy or sorafenib-based combination, patients must have received at least 14 days of sorafenib treatment with the lowest dosage of 400 mg per day.
* At least one measurable tumor, according to RECIST version 1.1, that has not been treated with any local procedure.
* ECOG performance status 0 or 1.
* Child-Pugh class A liver function.

Exclusion Criteria:

* Receiving concurrent anti-cancer therapy for HCC, which includes local therapy, chemotherapy, or other experimental therapy.
* Local treatment including radiotherapy (except palliative radiotherapy), percutaneous ethanol injection, radiofrequency ablation, transarterial embolization, or cryotherapy administered within 4 weeks prior to enrollment.
* History of HCC tumor rupture.
* Presence of brain or leptomeningeal metastases.
* Esophageal/gastric varices or active peptic ulcers that are considered to have high risk of bleeding.
* History of upper gastrointestinal bleeding within 1 year.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
disease stabilization | 8 weeks until tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Chiun Hsu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Shao YY, Chen BB, Ou DL, Lin ZZ, Hsu CH, Wang MJ, Cheng AL, Hsu C. Lenalidomide as second-line therapy for advanced hepatocellular carcinoma: exploration of biomarkers for treatment efficacy. Aliment Pharmacol Ther. 2017 Oct;46(8):722-730. doi: 10.1111/apt.14270. Epub 2017 Aug 17. PMID 28815645